CLINICAL TRIAL: NCT00004892
Title: Phase I GLIADEL and Continuous Infusion of Intravenous O6-Benzylguanine Trial in Patients With Recurrent Malignant Glioma
Brief Title: O6-Benzylguanine and Carmustine Implants in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067569; NABTT-9803; JHOC-NABTT-9803
Record Dates: First submitted 2000-03-07; First posted 2004-05-03 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult brain stem glioma; adult ependymoma; adult glioblastoma; adult oligodendroglioma; adult anaplastic astrocytoma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Ependymoma; Glioblastoma; Oligodendroglioma; Astrocytoma; Glioma; Gliosarcoma | interventions — O(6)-benzylguanine; Carmustine

INTERVENTIONS:
Drug: O6-benzylguanine
Drug: polifeprosan 20 with carmustine implant
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving drugs in different ways may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of O6-benzylguanine and implanted carmustine wafers in treating patients who have recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the dose of O6-benzylguanine that completely suppresses AGT levels in patients with recurrent malignant glioma. II. Evaluate the safety and tolerance of increasing duration for up to 2 weeks of continuously infused O6-benzylguanine at a dose that will completely suppress tumor AGT activity combined with intracranially implanted polifeprosan 20 with carmustine implants (Gliadel wafers) in this patient population.

OUTLINE: This is a dose escalation study of O6-benzylguanine (O6-BG). Patients in the first cohort receive O6-BG IV over 1 hour followed by continuous infusion of O6-BG for 2 days prior to surgery. Patients undergo surgical resection and receive up to 8 polifeprosan 20 with carmustine implants (Gliadel wafers) in the resected tumor cavity. Cohorts of 14 patients receive escalating doses of O6-BG until 11 out of 14 patients in a cohort have complete suppression of AGT levels. Once the dose of O6-BG that completely suppresses AGT has been established, subsequent patients receive O6-BG IV beginning at least 1 hour prior to surgery followed by the established continuous infusion dose beginning on the day of surgery. The infusion continues for up to 14 days postoperatively. Cohorts of 6-12 patients receive lengthened durations of continuous infusion O6-BG until the maximum tolerated dose (MTD) is determined or the length of the infusion reaches 14 days. The MTD is defined as the dose preceding that at which 3 of 6 or 5 of 12 patients experience dose limiting toxicities. Patients are followed at 3, 6, 9, and 12 months, and then until death.

PROJECTED ACCRUAL: A minimum of 38 patients will be accrued for this study over 9.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignant glioma determined from prior stereotactic biopsy or cytoreductive surgery for removal of a supratentorial brain tumor Unilateral supratentorial tumor, measuring at least 1 cm, as determined by CT scan or MRI No more than 1 focus of tumor and no tumor crossing the midline Surgical treatment indicated at baseline evaluation Received prior definitive (greater than 5,000 cGy) external beam radiotherapy more than 3 months ago Evidence of progression At time of tumor resection and Gliadel wafers implantation: Intraoperative pathological diagnosis on frozen section or squash preparation of malignant glioma OR Glioblastoma multiforme or anaplastic astrocytoma on permanent sections from a prior surgery and an intraoperative pathological diagnosis on frozen section or squash preparation of tumor, glioma, or malignant glioma (not necrosis)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: At least 60 days Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases no greater than 4 times upper limit of normal Renal: Creatinine no greater than 1.7 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception for 1 year after surgery No other concurrent significant life threatening disease No known hypersensitivity to nitrosoureas No other malignancy in past five years except curatively treated carcinoma in situ of the cervix or basal cell carcinoma of the skin

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered No other concurrent chemotherapy during first 56 days of study Endocrine therapy: No concurrent dexamethasone as an antiemetic Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-04

CONTACTS AND LOCATIONS:
Overall Officials: Jon Weingart, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (9):
- United States (9):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Result] Weingart J, Grossman SA, Carson KA, Fisher JD, Delaney SM, Rosenblum ML, Olivi A, Judy K, Tatter SB, Dolan ME. Phase I trial of polifeprosan 20 with carmustine implant plus continuous infusion of intravenous O6-benzylguanine in adults with recurrent malignant glioma: new approaches to brain tumor therapy CNS consortium trial. J Clin Oncol. 2007 Feb 1;25(4):399-404. doi: 10.1200/JCO.2006.06.6290. PMID 17264335